CLINICAL TRIAL: NCT05558475
Title: Path To Better Sleep + Virtual Coaching: The Effectiveness and Implementation of Internet-Based Self-Management Program for Insomnia in a Regional Healthcare System
Brief Title: The DigIT Trial: The Effectiveness and Implementation of a Coached Digital Insomnia Treatment Program in a Regional Healthcare System.
Acronym: DigIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 20-253
Record Dates: First submitted 2022-09-22; First posted 2022-09-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Insomnia Disorder
Keywords: Health Technology; Internet-based program; Self-management; Primary Care; Mental Health; Digital CBTi
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A pragmatic mixed-models hybrid type-2 effectiveness-implementation trial will be used. 1) the effectiveness of a bundled clinical intervention: Digital CBTi plus Virtual Coaching Support (Digital CBTi with Coaching); and 2) a scalable implementation strategy for Digital CBTi with Coaching (REP-DI). The setting will be five healthcare systems within VISN 1: VA Maine, VA Central Western Massachusetts, VA White River Junction, VA Connecticut, and the Manchester VA. Interested and appropriate participants will undergo patient-level 1:1 stratified randomization to receive either Digital CBTi with Coaching or Digital CBTi+ Contact (control). All organizations will receive implementation activities and all participants will receive usual medical care.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital CBTi with Coaching (Experimental): Virtual Coaching integrated with Digital CBTI. Includes initial enrollment contact, onboarding call, and two follow-up support calls. The coach will be available as resource for technical and other support.
  Interventions: Behavioral: Virtual Coaching
- Digital CBTi without Coaching (+ initial contact) (No Intervention): The control will be an enhanced treatment as usual condition where participants will receive: 1) provider referral to Digital CBTi; 2) initial enrollment contact and 3) NO virtual coaching contacts. If subjects have a question or need technical support, they will be instructed to contact study staff for assistance.

INTERVENTIONS:
Behavioral: Virtual Coaching — The core coaching components are motivational support, clinical health education, and technical support. The specific objectives are: support PTBS engagement, foster subsequent treatment adherence, ensure appropriate implementation of guidelines for Sleep Restriction Therapy and Stimulus Control, identify and triage PTBS candidates who are not appropriate or need more intensive treatments, and provide PTBS course technical support.
  Arms: Digital CBTi with Coaching

SUMMARY:
The study will evaluate the effectiveness and implementation of a Virtual Coaching Intervention to enhance use of a digital intervention delivering cognitive behavioral therapy for insomnia (digital CBTi) at primarily rural VISN 1 facilities. The digital CBTi program was developed by VA specifically for Veterans. The Digital CBTi program contains the core elements of CBTi (sleep restriction, stimulus control, etc.) and matches the form of commercial digital CBTi programs, but is publicly available, currently in use in VA, and includes unique activities such as Veteran videos and various sleep diary options. A virtual coaching intervention, where a coach based in VA Connecticut will provide telephone coaching support to Veterans referred to Digital CBTi across VISN 1 sites, will increase engagement and adherence while fostering improved clinical outcomes. The investigators have hypothesized that Veterans randomized to Digital CBTi with Coaching will report greater improvement in insomnia severity and sleep parameters compared to Digital CBTi plus Contact (an enhanced treatment as usual control that provides an initial contact but NO coaching). The strategy used to implement Digital CBTi with Coaching will result in adequate Reach among Veterans (operationalized as 5 progressive levels of Veteran engagement in Digital CBTi) and Adoption among providers (2 progressive levels of provider engagement). A three-part formative evaluation of implementation (pre-implementation, active implementation, maintenance) consisting of interviews with Veterans, providers, and staff will optimize implementation in real time by tailoring implementation strategy elements to specific contexts.

DETAILED DESCRIPTION:
Background:

As many as 1.8 million individuals using VA services meet criteria for insomnia disorder, a condition associated with suicide, poor functioning, and medical as well as mental health disorders. Cognitive Behavioral Therapy for insomnia (CBTi) is the gold-standard treatment. However, only a small fraction of Veterans receive CBTi due to a host of barriers, including lack of providers, travel, scheduling and stigma, which are particularly relevant to those using rural and low-resourced treatment settings. A digital intervention delivering CBTi has been developed by VA specifically for Veterans. PTBS, enhanced by personal coaching, may mitigate barriers to CBTi by enabling self-management beyond clinic walls.

Significance:

Current Digital CBTi dissemination practices consist of inadequate messaging, poor integration into clinical workflow, and the absence of personal support. Preliminary data indicate that while Digital CBTi has increased access to CBTi, only an estimated 0.8% of Veterans with insomnia disorder have visited the Digital CBTi site. To address these gaps, (1) coaching must be integrated with Digital CBTi (Digital CBTi with Coaching) to increase engagement/adherence and (2) Digital CBTi with Coaching must be embedded in current VA care practices using a scalable implementation strategy for digital interventions. Although other low impact or digital interventions for insomnia are in use by VA, the prevalence of insomnia far outweighs VA's capacity to deliver gold-standard treatment through any single modality. An array of treatment options is needed. Moreover, Digital CBTi coaching delivered through a hub-and-spoke model is a scalable approach to MISSION Act directives mandating evidence-based in rural areas.

Innovation and Impact:

The program is the first digital CBTi designed for Veterans. Digital CBTi is open access and meets stringent VA information security requirements. Coaching integrated into Digital CBTi will increase engagement and adherence. A hub-and-spoke model of coaching limits reliance on local facility resources. A scalable implementation strategy for digital interventions, optimized during an HSR&D career development award, will be used. The VISN 1 clinical trials network will allow access to a rural Veteran population and provide research coordination resources.

Specific Aims:

1. [Establish effectiveness of Digital CBTi with Coaching when implemented in rural-facing VISN 1 facilities] H1: Veterans randomized to Digital CBTi with Coaching will report greater improvement in insomnia severity (primary) and sleep parameters (secondary) compared to [Digital CBTi+ Contact (an enhanced treatment as usual control)]
2. Evaluate the quantitative outcomes of REP-DI, the strategy used to embed Digital CBTi with Coaching in VA care. H2: REP-DI will result in adequate Reach among Veterans, Adoption among providers, and Maintenance.
3. Conduct a 3-part (pre-implementation, active implementation, maintenance) formative evaluation of implementation. Interviews with Veterans, providers, and staff will be informed by constructs from the Consolidated Framework for Implementation Research (CFIR). Data will optimize implementation in real time by tailoring implementation strategy elements to specific contexts.

Methodology:

A pragmatic hybrid type-2 effectiveness/implementation mixed-methods trial will be used. Outpatients with insomnia disorder will be referred by VISN 1 providers and randomized to either Digital CBTi with Coaching or Digital CBTi with contact. The implementation strategy will be REP-DI, a scalable and resource efficient strategy for implementing digital interventions. REP-DI will include provider training and augmentation of site referral processes, among other activities, to support PTBS implementation. Outcomes will be evaluated according to the RE-AIM framework. Digital CBTi with Coaching effectiveness outcomes include insomnia severity (primary), sleep parameters, fatigue, mood, sedative-hypnotic use, and other measures collected at baseline, 8 weeks, and 6 months. REP-DI quantitative implementation outcomes will include progressive levels of Reach, Adoption, and Maintenance evaluated at patient and provider/staff levels. A 3-part formative evaluation of implementation and implementation strategy optimization process will identify patient and provider/staff determinants through qualitative analysis of semi-structured interviews.

Next Steps/Implementation:

Digital CBTi with Coaching can be implemented across VA using REP-DI by the National Center for Health Promotion and Disease Prevention and secondary VA partners such as the Offices of Rural Health and Connected Care.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who meet the ICSD-3 Insomnia disorder diagnostic criteria,
* have an interest in digital CBTi, and
* have basic technology literacy.

Exclusion Criteria:

* Nighttime or Rotating Shift Work within the last 6 Months,
* Disorders: Psychotic DO; Bipolar DO;
* Dementia;
* moderate Cognitive Impairment;
* Epilepsy;
* Seizure DO,
* Severe OSA: untreated or treatment non-adherence,
* Current Exposure Therapy for PTSD

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | change from baseline to 10 weeks
  The ISI is the standard for self-reported insomnia symptoms. The ISI is a 7-item questionnaire (5-point Likert scale, total score ranges from 0-28) providing a global measure of perceived insomnia severity. The ISI has adequate psychometric properties and has been validated against sleep diary and polysomnographic measures of sleep.
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Insomnia Severity Index (ISI) | change from baseline to 6 months
  The ISI is the standard for self-reported insomnia symptoms. The ISI is a 7-item questionnaire (5-point Likert scale, total score ranges from 0-28) providing a global measure of perceived insomnia severity. The ISI has adequate psychometric properties and has been validated against sleep diary and polysomnographic measures of sleep.
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)

SECONDARY OUTCOMES:
Sleep Onset Latency (SOL) | change from baseline to 10 weeks
  Sleep onset latency (SOL) is the length of time that it takes to accomplish the transition from full wakefulness to sleep. It is measured in minutes where high number means longer time and low number means shorter time to fall asleep.
Sleep Onset Latency (SOL) | change from baseline to 6 months
  Sleep onset latency (SOL) is the length of time that it takes to accomplish the transition from full wakefulness to sleep. It is measured in minutes where high number means longer time and low number means shorter time to fall asleep.
Sleep Efficiency (SE) | change from baseline to 10 weeks
  Sleep efficiency (SE), commonly defined as the ratio of total sleep time to time in bed. It is given as a percentage where high percentage indicates normal/healthy SE (ex. 80-90%) while low percentage indicates low SE.
Sleep Efficiency (SE) | change from baseline to 6 months
  Sleep efficiency (SE), commonly defined as the ratio of total sleep time to time in bed. It is given as a percentage where high percentage indicates normal/healthy SE (ex. 80-90%) while low percentage indicates low SE.
Wake After Sleep Onset (WASO) | change from baseline to 10 weeks
  WASO (wake after sleep onset) is defined as an unwanted wake or waking period after sleep onset. By definition, sleep must continue after the wake in order for it to count as a WASO. WASO is measures in minutes where high number means longer time awake and low number means shorter time awake after sleep onset.
Wake After Sleep Onset (WASO) | change from baseline to 6 months
  WASO (wake after sleep onset) is defined as an unwanted wake or waking period after sleep onset. By definition, sleep must continue after the wake in order for it to count as a WASO. WASO is measures in minutes where high number means longer time awake and low number means shorter time awake after sleep onset.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hermes, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT; Christi S. Ulmer, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (5):
- United States (5):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Maine VA Medical Center, Augusta, ME, Augusta, Maine
  - VA Central Western Massachusetts Healthcare System, Leeds, MA, Leeds, Massachusetts
  - Manchester VA Medical Center, Manchester, NH, Manchester, New Hampshire
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-08-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT05558475/ICF_000.pdf